CLINICAL TRIAL: NCT04753580
Title: Sampling of Human Microbiota in Order to Test, on a Mouse Model, Individualized Intervention Strategies During Aging
Acronym: FRAGIBIOTE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Unite de Nutrition Humaine UMR 1019- INRAE (Unknown); Unite MetaGenoPolis INRAE (Unknown); France MICALIS Equipe ProbiHote UMR INRAE (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RBHP 2020 PICKERING 3; 2020-A02978-31 (Other: 2020-A02978-31)
Record Dates: First submitted 2021-02-11; First posted 2021-02-15 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-07

CONDITIONS: Healthy Volunteers; Frail Volunteers
Keywords: Genetic; Elderly; Microbiota

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group 1 (Experimental): healthy adult 20-35 years old
  Interventions: Genetic: Stool collection
- group 2 (Experimental): healthy elderly 65+ years old
  Interventions: Genetic: Stool collection
- group 3 (Experimental): Frail elderly 65+ years old
  Interventions: Genetic: Stool collection

INTERVENTIONS:
Genetic: Stool collection — The volunteer will receive the stool collection kit as well as the procedure to follow for this collection.
  Treatment of stool after collection:
  The stool will be treated according to the following two procedures:
  i) part of the stool will be sequenced and will be stored as quickly as possible (4 hours maximum) at -80 ° C, 3 separate aliquots of 1 g; ii) the other part will be intended for implantation in rats and must be homogenized in a final concentration of 20% glycerol (2 hours maximum) and then stored at -80 ° C, 3 aliquots of 1 g.

SUMMARY:
Human microbial flora transfer studies in rodent models have clearly identified that age-associated microbiota dysbiosis can play a decisive role with respect to pathologies or complications linked to aging: increased intestinal permeability, in place of systemic inflammation, dysfunction of immune cells and insulin resistance.

This trial therefore aims to validate the process of ex vivo transfer to the rat of human microbiota selected from three categories of male individuals: young adults, healthy older adults and frail older adults, with the evaluation of the bacterial population of stool by analysis of the 16S rRNA gene.

DETAILED DESCRIPTION:
This is a pilot study to validate a process of ex vivo stool transfer from humans to rats. Single-center intervention research with minimal risks and constraints.

Exploration of the bacterial composition of the intestinal microbiota in healthy adult volunteers, healthy elderly and frail elderly. The evaluation of the bacterial population of the stool will be done by analysis of the 16S rRNA gene.

The secondary objectives will evaluate the muscular functional abilities the body composition measurement, at Day 0 (visit 2) and the inflammatory status at Day -7 (visit 1).

Seconds parameters are the following :

seated, standing, walking, and direction changes, a balance test, a walking speed test and a chair lift test, the maximum voluntary force of manual gripping, the maximum muscle strength of the quadriceps and the level of autonomy

This protocol includes 3 visits :

* Visit 1 : Day -7 (allowed until Day-14) = inclusion
* Visit 2 : Day 0 = tests and questionnaires
* Visit 3 : Day +7 (allowed from Day+1) = stool collect

ELIGIBILITY:
Inclusion Criteria:

* Volunteer over the age 18,
* More than 50 kg and having a Body Mass Index (BMI) between 18 and 30 kg / m2 (inclusive),
* Subject aged between 20 and 35 years inclusive ("healthy adult" group, or 65 years (inclusive) and over ("healthy elderly" and "frail elderly" groups),
* Score of the Short Emergency Geriatric Assesment grid (SEGA - A) strictly less than 8 (see appendix 1) ("healthy adult" and "healthy elderly" groups), or greater than or equal to 8 ("frail elderly" group),
* Subject capable of giving informed consent to participate in the research,
* Subject having an affiliation to the French Social Security system.

Exclusion Criteria:

Healthy adult group and Healthy elderly group:

* Subject presenting an acute pathology (unstable pathology), a life expectancy of <3 months or major neuro-cognitive disorders,
* treated with antibiotic therapy 3 months before the start of the protocol,
* in the impossibility of carrying out the planned functionality tests,
* carrier of Pacemaker or implantable defibrillator,
* with renal insufficiency (clearance <50 ml / min according to the CKD-EPI formula),
* presenting an untreated metabolic syndrome (presenting 3 of the 5 following criteria: waist circumference greater than 94 cm, blood triglyceride level greater than 1.7 mmol / l, blood pressure greater than or equal to 130 mm Hg / 85 mm Hg, cholesterol level (HDL) less than 1.0 mmol / l, fasting blood glucose greater than or equal to 5.6 mmol / l),
* suffering from diabetes (even treated),
* during a slimming diet,
* during treatment with chemotherapy,
* with gastrointestinal pathology,
* with intolerance (milk, lactose, gluten ...) or a diet other than omnivorous (vegetarians, vegans, vegans),
* smoking more than 4 cigarettes / day,
* drinking more than 2 glasses of alcohol per day,
* refusing not to smoke, vape or remove a nicotine patch the morning of the samples,
* having a biological assessment judged by the investigator to be incompatible with the test,
* having a medical and / or surgical history judged by the investigator to be incompatible with the test,
* having drug treatments or nutritional supplements judged by the investigator to be incompatible with the test, (see detail in 8.5)
* having cooperation and understanding that does not allow strict compliance with the conditions set out in the protocol,
* participating in another clinical trial, or being in an exclusion period, or having received a total amount of compensation greater than 4500 euros over the 12 months preceding the start of the trial,
* benefiting from a legal protection measure (curatorship, guardianship, safeguard of justice),
* refusing to participate in the study.

Fragile elderly group:

Same non-inclusion criteria as above except modification on 2 criteria:

* Renal failure (clearance <30 ml / min according to the CKD-EPI formula)
* No restriction on the parameters defining the metabolic syndrome unless the subject has treated insulin-dependent diabetes.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2022-09-14 (Actual); Study Completion 2022-09-14 (Actual)

PRIMARY OUTCOMES:
Evaluation of the bacterial population of the stool by analysis of the 16S rRNA gene | Day +7
  Random metagenomic sequencing. The DNA sequences obtained will be aligned with catalogs of genes and microbial species representative of the gut microbiota to obtain a detailed microbial and functional profile (catalog of 10.4 million genes and ~ 2000 intestinal microbial species)

SECONDARY OUTCOMES:
Measurement of muscular functional aptitudes with the Get up and Go muscular test scale | Day 0
  Test that assesses seated, standing, walking and changes of direction transfers. This is a simple validated field test modified secondarily by adding the measured time. The subject is seated on a chair with armrests, placed in front of a wall 3 meters away. The subject should stand up, remain standing, walk to the wall, turn around without touching the wall, return to the seat, walk around it and sit down again. The rating is carried out with a scale rated from 1 to 5: 1 - no instability ; 2 - very slightly abnormal (slow execution) ; 3 - moderately abnormal (hesitation, compensatory movements) ; 4 - abnormal (the patient trips) ; 5 - very abnormal (permanent risk of falling).
Measurement of muscular functional aptitudes with the Short Physical Performance Battery (SPPB) score | Day 0
  This test includes a balance test, a walking speed test and a chair lift test. It makes it possible to assess the physical performance of an individual. Adding up the scores for all tests provides an overall performance score. A score of less than 8 is an indicator of the risk of sarcopenia (or age-related muscular dystrophy)
Evaluation of the the maximum voluntary force of manual gripping. | Day 0
  Measurement (in Newton) carried out on the dominant limb in a seated position, elbow resting on a table, with a Jamard dynamometer. The subject must make a gripping movement as hard as possible. Three reproducible measurements (+/- 10%) will be taken at 1 minute intervals and the highest value will be retained.
Evaluation of the voluntary level of autonomy with Functional Independence Measure (FIM) questionnaire | Day 0
  This test includes 18 items that assess a person's level of autonomy in their daily activities. Motor skills are measured by 13 tasks which are grouped under 4 categories of activities:
  Cognitive abilities are measured by 5 tasks which are grouped under 2 categories of activities:
Measurement of the distance travelled in 6 minutes with the 6-minute walk test | Day 0
  6-minute walk test performed according to ATS recommendations. Measurement of the distance travelled in 6 minutes in a lane of 30 meters by the subject with collection of basic parameters (heart rate).
Fat mass ratio determination | Day 0
  The percentage of fat mass (%) (body composition) will be determined on each participant using a multi-frequency bioelectrical Impedance Analyzer.
Lean mass ratio determination | Day 0
  The percentage of lean mass (%) (body composition) will be determined on each participant using a multi-frequency bioelectrical Impedance Analyzer.
Water mass ratio determination | Day 0
  The percentage of water (%) (body composition) will be determined using a multi-frequency bioelectrical Impedance Analyzer.
Evaluation of the participant nutritional state with Mini Nutritional Assessment (MNA) | Day -7
  The Mini Nutritional Assessment is structured in 18 questions grouped in four rubrics (anthropometry, general status, dietary habits, and self-perceived health and nutrition states). It allows grading the nutritional status according to defined thresholds: scores above 24 = good status; scores 23.5-17 = risk of malnutrition; scores below 17 = malnutrition.
Evaluation of the participant cognitive state with Mini Mental State Examination (MMSE) | Day -7
  The Mini Mental State Examination is structured in 30 questions grouped in six rubrics (orientation, registration, attention and calculation, memory, language, and copying). It allows the screening of cognitive impairments.
Plasma glucose dosage | Day -7
  Determination of glucose plasma concentration (mmol/L) (a metabolic parameter).
Plasma creatinine dosage | Day -7
  Determination of creatinine plasma concentration (µmol/L) (a metabolic parameter).
Creatinine clearance | Day -7
  Determination of the creatinine clearance (ml/min) (a metabolic parameter).
Plasma albumin dosage | Day -7
  Description: Determination of albumin plasma concentration (a metabolic parameter).
Plasma total cholesterol dosage | Day -7
  Determination of total cholesterol plasma concentration (mmol/L) (a metabolic parameter).
Plasma High Density Lipoprotein cholesterol (HDL-chol) dosage | Day -7
  Description: Determination of HDL-chol plasma concentration (mmol/L) (a metabolic parameter).
Plasma triglycerides dosage | Day -7
  Determination of triglycerides concentration (mmol/L) (a metabolic parameter).
Plasma liver enzymes (AST/ALT/GGT) dosage | Day -7
  Determination of liver enzymes concentration (U/L) (a metabolic parameter).
Plasma phosphatase alkaline dosage | Day -7
  Determination phosphatase alkaline concentration (U/100mL) (a metabolic parameter).
Plasma C-reactive protein dosage | Day -7
  Determination C-reactive protein concentration (a metabolic parameter).
Complete blood count (CBC) | Day -7
  Determination of the number of erythrocytes (millions/mm3), leukocytes (mm3/1000), platelets (mm3/1000), the hematocrit rate (%), the hemoglobin rate (g/100ml), the mean corpuscular hemoglobin (pg), mean corpuscular volume (µ3), mean corpuscular hemoglobin concentration (%)
Dosage of TNF-alpha allowing assessment of inflammatory status | Day -7
  Determination of TNF-alpha plasma concentration (pg/ml)
Dosage of IL1 allowing assessment of inflammatory status | Day -7
  Determination of IL-1 plasma concentration (pg/ml)
Dosage of IL6 allowing assessment of inflammatory status | Day -7
  Determination of IL-6 plasma concentration (pg/ml)
Dosage of MCP1 allowing assessment of inflammatory status | Day -7
  Determination of MCP1 plasma concentration (pg/ml)
Dosage of IL10 allowing assessment of inflammatory status | Day -7
  Determination of IL10 plasma concentration (pg/ml)
Dosage of LPS-binding protein allowing assessment of inflammatory status | Day -7
  Determination of LPS-binding protein plasma concentration (ng/ml)
Dosage of sDC14 allowing assessment of inflammatory status | Day -7
  Determination of sDC14 plasma concentration (ng/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Gisèle PICKERING, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU, Clermont-Ferrand, France